CLINICAL TRIAL: NCT05475353
Title: The Effects of Ergonomics Awareness Education and Exercise on Physical Activity, Quality of Life, and Musculoskeletal Discomfort in Remote Workers
Brief Title: The Effects of Ergonomics Awareness Education and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Kültür University (Other)
Responsible Party: Principal Investigator, Halenur Evrendilek, Research Assistant, Istanbul Kültür University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2/2021.K-20
Record Dates: First submitted 2022-07-23; First posted 2022-07-26 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2022-07

CONDITIONS: Ergonomics; Telerehabilitation; Musculoskeletal System Disorder; Quality of Life
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asyncronized Exercise Group (Active Comparator): - Ergonomics awareness education and exercise suggestions
  Interventions: Behavioral: Asyncronized Exercise
- Syncronized Exercise Group (Experimental): - Ergonomics awareness education and than 6 weeks online supervised exercise training
  Interventions: Procedure: Syncronized Exercise

INTERVENTIONS:
Behavioral: Asyncronized Exercise — This group will be informed about ergonomics and protective exercises for the musculoskeletal system with an online seminar.
  Arms: Asyncronized Exercise Group
Procedure: Syncronized Exercise — This group will be informed about ergonomics and protective exercises for the musculoskeletal system with an online seminar. Then, participants will complete the 6 weeks of exercise training at an online video conference program two times a week under the physiotherapist's supervise.
  Arms: Syncronized Exercise Group

SUMMARY:
This study aims to determine the effects of asynchronous and synchronous exercises, which are added to ergonomics awareness education, on musculoskeletal disorders, physical activity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-45
* Working at home at least 5 hours a day
* Not having one or more diagnosed musculoskeletal disorders

Exclusion Criteria:

* Limited access to technology or not being able to actively use the technology
* Had musculoskeletal trauma or surgery
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Physical activty status | Baseline
  International Physical. Activity Questionnaire-short form
Physical activty status | 6 weeks
  International Physical. Activity Questionnaire-short form
Quality of life status | Baseline
  Short Form 36
Quality of life status | 6 weeks
  Short Form 36
Musculoskeletal Discomfort level | Baseline
  Cornell Musculoskeletal Discomfort Questionnaires: Higher scores indicate higher musculoskeletal discomfort.
Musculoskeletal Discomfort level | 6 weeks
  Cornell Musculoskeletal Discomfort Questionnaires: Higher scores indicate higher musculoskeletal discomfort.
Ergonomic risk level | Baseline
  Rapid Upper Limb Assesment: Higher scores indicate higher risk.
Ergonomic risk level | 6 weeks
  Rapid Upper Limb Assesment: Higher scores indicate higher risk.

CONTACTS AND LOCATIONS:
Overall Officials: Halenur Evrendilek, Res. Asst., Study Director — İstanbul Kültür University; Burcu Semin Akel, Prof. Dr., Study Director — İstanbul Kültür University
Locations (1):
- İstanbul Kültür Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No